CLINICAL TRIAL: NCT06175559
Title: Embedded Narrative in Interactive Game Design for Improving Medication Adherence of Schizophrenia：Exploratory Research
Brief Title: Embedded Narrative in Interactive Game Design for Improving Medication Adherence of Schizophrenia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: We have finished the first-stage study.
Sponsor: Zhu Dian (Other)
Responsible Party: Sponsor-Investigator, Zhu Dian, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Sjtu0002
Record Dates: First submitted 2023-12-08; First posted 2023-12-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia and Related Disorders; Medication Adherence; Mental Health Issue; Gamification
MeSH Terms: conditions — Schizophrenia; Medication Adherence | interventions — Research Design

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healing Town: Embedded Narrative in Interactive Game Design (Experimental): The game-based medication intervention game "Wanping Town" in this study employed a multidisciplinary participatory design approach rooted in narrative theory and behavioral psychology models. The game consists of two perspectives: narrative decision stories and cognitive games. The investigators initially employed participatory design methods to determine the plot and elements within the game, then embedded the conclusions into the therapeutic elements of the game.
  Interventions: Combination Product: Healing Town: Embedded Narrative in Interactive Game (Psycho-education Tool) Design

INTERVENTIONS:
Combination Product: Healing Town: Embedded Narrative in Interactive Game (Psycho-education Tool) Design — The narrative-based medication intervention game "Healing Town" in this study employed a multidisciplinary participatory design approach rooted in narrative theory and behavioral psychology models. The game consists of two perspectives: narrative decision stories and cognitive games. The investigators initially employed participatory design methods to determine the plot and elements within the game, then embedded the conclusions into the therapeutic elements of the game

SUMMARY:
This study explores the potential of an interactive narrative game to enhance medication adherence among stable schizophrenia patients. Employing participatory design methods, game's development and testing process actively involved patients and individuals closely connected to their daily lives. Artificial Intelligence-Generated Content (AIGC) facilitated swift iterations in game's visual style and content. During game therapy, patients are tasked with making decisions based on presented situations, which influence the course of the narrative.

DETAILED DESCRIPTION:
Our game design is inspired by Cognitive Behavioral Therapy (CBT), specifically the autonomic engagement and emotion regulation for the treatment of stable schizophrenic patients. This design aims to motivate patients to practice the basic principles of CBT in a virtual environment with the aim of producing positive psychological and behavioral changes in real life.

To ensure that the interactive design in the game can effectively promote cognitive reconstruction and emotional regulation in patients, the investigators used the following game interaction strategies:

1. Situational simulation: By simulating real-life situations, patients face challenges and make decisions in the game that are similar to those in real life, so as to train their cognitive and emotional regulation.
2. Immediate feedback: Provide patients with immediate feedback during the game so that they can understand the impact of their decisions on the outcome of the game, thus encouraging them to make more positive decisions in real life.
3. Role-imitation: Encourage patients to take an in-depth look at their thoughts and behaviors from a third-person perspective by having them take on the role of a therapy practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Stable Phase Schizophrenia
* on long-term medication
* medication adherence was problematic

Exclusion Criteria:

* Serious Schizophrenia
* Lack of basic cognitive abilities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | 10 minutes
  Medication Adherence - Morisky Medication Adherence Scale-8 (MMAS-8): This scale assesses medication adherence through 8 items, providing a comprehensive evaluation of adherence.
Medication Attitude | 10 minutes
  Medication Attitude - Drug Attitude Inventory (DAI) : This scale evaluates patients' attitudes toward medication, with higher scores indicating better attitudes.

SECONDARY OUTCOMES:
Game Experience | 10 minutes
  the In-Game Core Scale (iGEQ): a standardized tool used to measure a player's experience while playing a video game. It was developed by researchers to understand how players feel during gameplay, based on psychological and emotional factors.
Anxiety | 10 minutes
  Anxiety - Generalized Anxiety Disorder 7 (GAD-7) : This scale measures the level of anxiety in individuals, categorizing the severity into mild, moderate, and severe levels.
Depression | 10 minutes
  Depression - Patient Health Questionnaire-9 (PHQ-9): This scale assesses the severity of depressive symptoms, categorizing the level of depression from mild to severe.
Patients' Quality of Life | 10 minutes
  World Health Organization Quality of Life-BREF (WHOQOL-BREF) : This scale evaluates overall quality of life and health status, with a focus on physical, psychological, social, and environmental domains.
Social Functioning | 10 minutes
  Social Disability Screening Schedule (SDSS): This scale assesses the degree of social disability, with higher scores indicating more severe social dysfunction.
Clinical Symptoms | 10 minutes
  Clinical Symptoms - Brief Psychiatric Rating Scale (BPRS): This scale evaluates clinical symptoms across five factors, including anxiety-depression, lack of vitality, thought disturbances, activation, and hostile suspicion.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Liu, Prof, Study Director — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
You can contact the author to obtain data, including patient medication adherence data before and after the experiment, interview data, and questionnaire data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the article is accepted
Access Criteria: zhudian@sjtu.edu.cn

REFERENCES:
- [Derived] Liu Z, Zhu D, Zhang Z, Liu Y, Yang H, Chang F, Zhang W, Cai J. Effects of a narrative-based psychoeducational intervention on medication adherence in individuals with schizophrenia: a multicentre, parallel-group randomised controlled trial. EClinicalMedicine. 2025 Sep 4;88:103483. doi: 10.1016/j.eclinm.2025.103483. eCollection 2025 Oct. PMID 40979217